CLINICAL TRIAL: NCT04743349
Title: Steam Inhalations in Asymptomatic and Paucisymptomatic COVID-19 Patients
Brief Title: Steam Inhalations in COVID-19 Patients
Acronym: Steam-COVID
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties in enrollment
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Giancarlo la Marca, Pharm Sc, Meyer Children's Hospital IRCCS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Steam-COVID
Record Dates: First submitted 2021-02-05; First posted 2021-02-08 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Covid19; Coronavirus Infection; Coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): Steam inhalations
  Interventions: Procedure: Steam inhalations
- Control arm (No Intervention): No intervention

INTERVENTIONS:
Procedure: Steam inhalations — Exposure of airway mucosae to humidified steam through steam inhalation for at least 20 min (4 cycles of 5 min) daily, for 10 days.
  Arms: Experimental arm

SUMMARY:
The new coronavirus (SARS-CoV-2) causing COVID-19 is an RNA virus coated with a capsid and a peri-capsid crossed by glycoprotein structures. The external proteic structure, which attacks human cells, is a potential target to therapeutic interventions against virus replication in airways.

Since high temperature can cause irreversible denaturation of proteins and loss of SARS CoV and SARS CoV-2 infectivity was obtained after heating at 56 ◦C for 15 and 30 min in liquid environments respectively, we designed a protocol aimed at damaging SARS-CoV-2 capsid through steam inhalation cycles. Although the ominous consequences of COVID 19 infections has directed medical attention toward solidly established medical approaches, the European Pharmacopoeia VI edition also quotes steam inhalations as a procedure to treat of respiratory diseases.

Based on these suggestions we established a quasi-randomized clinical trial enrolling 200 asymptomatic or paucisymptomatic patients in whom rhino-pharyngeal-swab revealed a SARS-CoV-2 infection. The study protocol consisted of exposure of airway mucosae to humidified steam (pH 8 per NaHCO3 and hypertonic 15 g/L NaCl) through steam inhalation for at least 20 min (4 cycles of 5 min) daily, for 10 days.

The objective of the study is to reduce the viral shedding using steam inhalations.

ELIGIBILITY:
Inclusion Criteria:

* Adults with a SARS-CoV-2 positive molecular swab carried out in the previous 48 hours before the enrollement
* Adults with mild infection
* Adults with symptoms such as fever above 37 ° C, feeling bad, cold symptoms (cough, pharyngodynia, nasal congestion), headache, myalgia, diarrhea, anosmia, dysgeusia
* Adults without the above symptoms

Exclusion Criteria:

* Adults with dyspnea and/or dehydration and/or alterations in consciousness and/or sepsis.
* Subjects with severe asthma
* Subjects and with contraindications to treatment with steam inhalations
* Multi-allergic subjects
* Subjects unable to complete the protocol

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-06-06 (Actual)

PRIMARY OUTCOMES:
Reduction in viral shedding | From date of randomization until the date of first documented negativization from any cause assessed up to 9 months
  Difference / ratio between the percentage of subjects with negative swab 10 days after enrollment in the treated group and the percentage in the non-treated group.

SECONDARY OUTCOMES:
Clinical outcome | From date of randomization until the date of first documented clinical improvement from any cause assessed up to 9 months"
  Difference / ratio between the percentage of subjects with residual symptoms after 10 days of enrollment in the treated group and the percentage of subjects with residual symptoms after 10 days of enrollment in the untreated group (only for the subgroup of patients with severe symptoms).
Negativization rate | From date of randomization until the date of first documented negativization from any cause assessed up to 9 months
  Ratio between the incidence of the negativization rate (number of events / total person days) in the treated group and the incidence of the negativization rate in the untreated group.

OTHER OUTCOMES:
Viral load measurement | From date of randomization until the date of first documented negativization from any cause assessed up to 9 months
  Measurement expressed in pg / mL of the mean values of the viral load measured in the treated group compared to the untreated group at the different monitoring times

CONTACTS AND LOCATIONS:
Locations (1):
- Meyer Children's Hospital, Florence, Italy

IPD SHARING:
Plan to Share IPD: No